CLINICAL TRIAL: NCT04831801
Title: Trends in the Microbiome Profiles of Women With Urgency and Frequency Syndrome, With or Without Pelvic Pain?
Brief Title: OAB and the Microbiome
Status: Terminated | Type: Observational
Why Stopped: No longer with institution
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Laura Martin, Assistant Professor, University of Miami
Other Study IDs: 20201001
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Overactive Bladder; Urgency-frequency Syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female patients with overactive bladder (OAB): Patients with urgency and frequency syndrome with or without pelvic pain (Group A) will provide two urine samples. One urine sample is a clean catch and the other is a catheterized specimen. Both will be sent for analysis. A perineal swab will also be collect and analyzed for each patient.
- Female control patients without LUTS: Patients without LUTS (Group B) will provide two urine samples. One urine sample is a clean catch and the other is a catheterized specimen. Both will be sent for analysis. A perineal swab will also be collect and analyzed for each patient.

SUMMARY:
To determine differences in the urinary microbiomes, identified by polymerase change reaction (PCR) (UTIP™), of female patients with urgency and frequency syndrome with or without pelvic pain (Group A) compared to female controls without symptoms of lower urinary tract symptoms (LUTS) (Group B).

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o-90 y/o
* Able to consent
* Group A only: Urgency and Frequency Syndrome or OAB only. UDI-6 answer of "moderately" to "quite a bit" on questions 1 or 2.
* Group B only: Urinary Distress Inventory 6 (UDI-6) answer "not at all" or "somewhat" for questions 1 or 2.

Exclusion Criteria:

* Pregnant
* Pelvic radiation
* Urinary retention (>200 ml)
* Renal calculi
* Recurrent urinary tract infection (UTI) (2 in 6 months), or
* Current UTI
* Immunosuppressed or radiation history
* Neurologic disorder

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients with OAB and controls will be enrolled from University of Miami's or Holy Cross Hospital's female pelvic medicine and reconstructive surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Lactobacillus in samples. | Day 1
  Evaluation of urine and perineal samples by PCR.
Proportion of patients negative for repeat sequencing. | Day 1
  Evaluation of urine and perineal samples by PCR.
Proportion of patients with change in UDI-6 score | Up to 4 weeks
  UDI 6 question 1 and 2 has a total score from 0-6 with a high score indicating more distress. Proportion of patients with a decrease in score from baseline will be reported for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Martin, DO, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No